CLINICAL TRIAL: NCT07120165
Title: Effectiveness of Myopia Control Interventions : A Comparison of Myopia Control in European Children, Adolescents and Young Adults With Defocus Incorporated Multiple Segments (DIMS) and Highly Aspherical Lenslets (HAL) Spectacles, Atropine, Lenses and Combined Treatments
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1022025/CHUSTE
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Myopia
Keywords: Myopia; children; teenagers; atropine; lunettes; contact lenses; combinations
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Atropine 0.01%: Children or young adults with active myopia treated with ATROPINE 0.01% eye drops.
  Interventions: Other: Demographic data collection; Other: Ophthalmological history; Other: Ophthalmological data at each examination; Other: Potential adverse events
- DIMS/HAL: Children or young adults with active myopia treated with myopia control glasses.
  Interventions: Other: Demographic data collection; Other: Ophthalmological history; Other: Ophthalmological data at each examination; Other: Potential adverse events
- Various combined treatments: Children or young adults with active myopia treated with ATROPINE 0.01% eye drops or myopia control glasses or contact lenses, and their various combinations.
  Interventions: Other: Demographic data collection; Other: Ophthalmological history; Other: Ophthalmological data at each examination; Other: Potential adverse events

INTERVENTIONS:
Other: Demographic data collection — Demographic data collection: age, gender, level of education/study, time spent in near vision, sports practice, medical history
Other: Ophthalmological history — Ophthalmological history: age of myopia discovery, parental refraction, previous refractions, presence of a braking treatment
Other: Ophthalmological data at each examination — Ophthalmological data at each examination: visual acuity, subjective refraction, cycloplegia with SKIACOL, axial length.
Other: Potential adverse events — Potential adverse events: halos, photophobia, stinging, infections, etc.

SUMMARY:
The prevalence of myopia and its complications has risen considerably in recent decades, particularly among children and teenagers. This trend is also spreading in Europe, driven by the increase in screen time and the intensive use of new technologies and social media, particularly among the younger generation.

Several treatment options are available today, including pharmacological treatments with atropine eye drops, as well as optical myopia control systems in the form of glasses or contact lenses.

These different treatments have been used in clinical practice at Saint-Étienne University Hospital since 2017 for atropine, and more recently with the development of optical myopia control systems and their combinations.

Little clinical data has been published to date on these different treatment combinations in the French population.

The investigators would therefore like to set up a database to publish their results and share their experience.

ELIGIBILITY:
Inclusion Criteria:

* Children or young adults with active myopia treated with ATROPINE 0.01% eye drops or myopia control glasses or contact lenses, and their various combinations
* patient affiliated with a social security organization
* agreement of both parents or the patient if adult

Exclusion Criteria:

- non compliance with treatment

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children or young adults with active myopia treated with ATROPINE 0.01% eye drops or myopia control glasses or contact lenses, and their various combinations will be included.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Database of active treatments for myopia | Month 5
  Database established with data from children or young adults with active myopia treated with ATROPINE 0.01% eye drops or myopia control spectacles or contact lenses, and their various combinations.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Caroline TRONE, Md, Principal Investigator — CHU de Saint-Étienne
Locations (1):
- CHU de Saint-Étienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No